CLINICAL TRIAL: NCT00176579
Title: Assessing Bone Mineral Density as a Risk Factor for Early Clinically Significant Prostate Cancer
Brief Title: Bone Mineral Density and Cancer Recurrence in Patients With Early Stage Prostate Cancer
Status: Completed | Type: Observational
Sponsor: University of Medicine and Dentistry of New Jersey (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Stephen Marcella, UMDNJ/CINJ
Organization: Rutgers, The State University of New Jersey (Other)
Other Study IDs: CDR0000539677; P30CA072720 (NIH); CINJ-5004; CINJ-4375
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2011-08-12 (Estimated); Status verified 2011-08

CONDITIONS: Osteoporosis; Prostate Cancer
Keywords: osteoporosis; stage I prostate cancer
MeSH Terms: conditions — Osteoporosis; Prostatic Neoplasms | interventions — Absorptiometry, Photon

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: dual x-ray absorptiometry — Dual x-ray absortiometry by densitometer will be performed to measure bone mineral density

SUMMARY:
RATIONALE: Measuring bone mineral density may help doctors predict whether prostate cancer will come back. It may also help the study of prostate cancer in the future.

PURPOSE: This clinical trial is studying whether bone mineral density affects cancer recurrence in patients with early stage prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine bone mineral density (BMD) in patients with clinically significant early stage prostate cancer.
* Determine whether patients who have a higher level of BMD and have had a radical prostatectomy for cure are less likely to have an early relapse (i.e., less than 3 years) than those patients with a low level of BMD.

OUTLINE: This is a case-controlled study followed by a prospective, longitudinal, cohort study.

Patients undergo bone mineral density (BMD) measurements by dual-energy x-ray absorptiometry with a densitometer. Posteroanterior measurements of the total hip are also recorded.

Patients also undergo blood collection to examine markers that provide evidence of systemic disease.

Patients are followed every 6 months for 3 years.

PROJECTED ACCRUAL: A total of 40 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Biopsy-confirmed early stage prostate cancer

  * Disease localized within the capsule
  * No evidence of regional or distant spread (i.e., T1-2, N0, M0 disease)
  * A cohort of patients must have undergone a prior radical prostatectomy
* Prostate specific antigen < 12 ng/mL
* Gleason score ≥ 6

PATIENT CHARACTERISTICS:

* Creatinine clearance ≤ 2.0 mg/dL
* No Paget's disease
* No hyperthyroidism or hypothyroidism
* No Cushing's disease
* No chronic liver disease
* No major health problems that would cause a significant reduction in mobility or activities of daily living

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior bisphosphonates, thyroxin, or calcitonin
* No prior agents that suppress PSA levels (e.g., finasteride)
* No prior androgen or estrogen therapy
* More than 12 months since prior glucocorticoids
* More than 12 months since prior herbal supplements that are known to lower PSA levels

Ages: 50 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will be recruited from urologists' offices and the oncological practices of CINJ. This will be done by verbal communication through the office staff and with the distribution of a brochure briefly describing the study. If a person is interested, he will be given information that briefly describes the study and his name will be taken down. A research assistant will call him and set up a meeting, preferably at the same time he is scheduled to see his physician. At that meeting, a research assistant will go over the consent form with him and cover all questions concerning the study. Eligibility (based on history) will also be verified at this meeting. If he wishes to participate, he will be instructed to sign the consent and an appointment for the blood tests and DXA scan will be arranged.
Sampling Method: Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2003-06; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Bone mineral density | Baseline
  DXA scan will be done after patient signs consent and eligibilty is confirmed
Prostate Specific Antigen | Baseline, every 6 months for 3 years
  PSA will be measured to look for biochemical recurrence of prostate cancer

CONTACTS AND LOCATIONS:
Overall Officials: Stephen W. Marcella, MD, MPH, Principal Investigator — Rutgers Cancer Institute of New Jersey
Locations (1):
- Cancer Institute of New Jersey at UMDNJ - Robert Wood Johnson Medical School, New Brunswick, New Jersey, United States

REFERENCES:
- See also: Clinical trial summary from Clinicaltrials.gov website — http://clinicaltrials.gov/ct2/show/NCT00176579